CLINICAL TRIAL: NCT02354677
Title: Repair, Remodeling and Regeneration of the Bronchial Epithelium of COPD Patients
Acronym: RRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9244; 2013-A01405-40 (Other: RCB number)
Record Dates: First submitted 2015-01-12; First posted 2015-02-03 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2018-05

CONDITIONS: Heathy Volunteers; Smokers; COPD
Keywords: Bronchial epithelium; COPD; Repair; Remodelling; Club Cells
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heathy volunteers, smokers and COPD (Experimental)
  Interventions: Other: In vitro experiments on bronchial epithelial cells

INTERVENTIONS:
Other: In vitro experiments on bronchial epithelial cells

SUMMARY:
COPD is characterized by exagerated decline FEV1 related to obstructive non reversible airflow. This could be the consequence of structural changes and inflammatory pattern of the bronchial wall. Lesions could lead to normal but also abnormal remodeling specially in COPD including a decrease in Club cells number and function.There is no treatment actually available targeted to a normal repair of the epithelium. The objective of this work is to identify potential targets for reprograming bronchial epithelial cells I order to achieve a good repair.

ELIGIBILITY:
Inclusion Criteria:

COPD - Smokers or ex smokers > 30p/yr

* FEV1/FVC < 0.7
* With a fibroscopy prescription

Smokers - Smokers or ex smokers > 30p/yr

* FEV1/FVC > 0.7
* With a fibroscopy prescription

Controls - age superior or equal to 18

* no smoker (for 5 years)
* with a fibroscopy prescription

Exclusion Criteria:

* Xylocaine hypersensibility
* Porphyria
* severe hepatic failure
* Epilepsy
* Severe cardiac failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Full recovery one day after injury (yes / no) proportion of cells showing the repair, remodeling or regeneration of the epithelium (ciliated cells, mucus cells, Clara cells) in culture in air-liquid interface in the three groups | 1 day
  The study will be judged on the proportion of cells showing the repair, remodeling or regeneration of the epithelium (ciliated cells, mucus cells, Clara cells) in culture in air-liquid interface in the three groups.

SECONDARY OUTCOMES:
Measurement of apoptosis and inflammation (IL8) | 24 months
  Determine the molecular mechanisms and deleterious cell leading to poor repair of the epithelium in patients with COPD
Measure the effect of the CC10 protein secreted by Clara cells on the repair of the bronchial epithelium. | 24 months
  Measuring the reprogramming of the epithelium of COPD patients to a control-type epithelium

CONTACTS AND LOCATIONS:
Overall Officials: BOURDIN Aranud, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Pneumology Department, Montpellier, France